CLINICAL TRIAL: NCT05501158
Title: CYP2D6 Genotypes and Breast Cancer Clinical Outcomes in the Indonesian Population (Pengaruh Genotipe CYP2D6 Terhadap Efektivitas Penggunaan Tamoksifen Untuk Pasien Kanker Payudara ER+ Pada Populasi Indonesia)
Brief Title: CYP2D6 Genotypes and Breast Cancer Clinical Outcomes in the Indonesian Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nalagenetics Pte Ltd (Industry)
Collaborators: SJH Initiatives (Unknown); Indonesia University (Other); MRCCC Siloam Hospitals Semanggi (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-TMS-02-20201012
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study involving the breast cancer patients who participated in our previous study. Patients who are recommended to adjust their tamoxifen dosage to 40 mg and remain on tamoxifen 20 mg will be all followed up for 3 years to evaluate the clinical outcomes and medication side effects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose adjustment of tamoxifen (Experimental): Following the CPIC guidelines, those identified as Poor Metabolizers (PMs) and Intermediate Metabolizers (IMs) from our previous study are recommended to adjust their tamoxifen dosage to 40 mg per day.
  Interventions: Drug: Tamoxifen
- Standard dose of tamoxifen (No Intervention): Those identified as Normal Metabolizers (NMs) from our previous study remain on tamoxifen 20 mg per day.

INTERVENTIONS:
Drug: Tamoxifen — Suggesting an increase in the dose of tamoxifen to those who have suboptimum level of endoxifen due to their genetic variations
  Arms: Dose adjustment of tamoxifen

SUMMARY:
The utilization of tamoxifen is considerably high in Indonesia, with about 170,000 tamoxifen prescriptions filed in 2015. It is metabolized by the enzyme CYP2D6, resulting in its active metabolite, endoxifen, which has been proven to be effective in the prevention and treatment of breast cancer.

Studies showed the CYP2D6 gene has more than 100 variants; some of which are linked with reduced drug activity, while others do not have any pathological implications. The metabolizer profile of these variants is generally grouped into Ultra-rapid, Normal, Intermediate, and Poor Metabolizers (UM, NM, IM, and PM, respectively). In our previous study (NCT04312347), the investigators recruited 150 breast cancer patients who were taking adjusted dose of tamoxifen daily based on their CYP2D6 phenotype. Although the investigators have measured the endoxifen level of the patients with adjusted treatment, the clinical outcomes of the study are not yet conclusive.

ELIGIBILITY:
Inclusion Criteria:

1. female
2. diagnosed with ER+ breast cancer
3. have been genotyped and classified as PM and IM in the previous study
4. are recommended by doctor to take tamoxifen 40 mg according to their metabolizer profile
5. have finished the definitive therapy course (surgery, chemotherapy, or radiotherapy).

Exclusion Criteria:

1. have other primary cancer aside from breast cancer.
2. those with residual tumor cells/have experienced second primary breast tumor.
3. patients who are recommended by doctor to switch to aromatase inhibitors (AI)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival rate | 3 year
  The percentage of study participants who are still alive by the end of this study after being diagnosed with breast cancer
Progression Survival rate | 3 year
  The percentage of study participants who live with the disease but the disease does not get worse by the end of this study

OTHER OUTCOMES:
Long-term side effects of tamoxifen | 3 year
  Long-term side effects of tamoxifen, including heartburn, thromboembolic event, endometrial hyperplasia and uterine cancer, will also be monitored and documented using the Adverse Drug Reaction (ADR) reporting form provided by the Indonesian National Agency of Drug and Food Control.

CONTACTS AND LOCATIONS:
Overall Officials: Baitha Maggadani, MPharm, Study Chair — Fakultas Farmasi Universitas Indonesia; Arief Winata, MD, Study Chair — MRCCC Siloam Hospitals Semanggi; Samuel Haryono, MD, PhD, Principal Investigator — SJH Innitiatives; Fatma Aldila, PharmD, Study Chair — Nalagenetics Pte Ltd
Locations (1):
- MRCCC Siloam Hospitals Semanggi, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braal CL, Jager A, Hoop EO, Westenberg JD, Lommen KMWT, de Bruijn P, Vastbinder MB, van Rossum-Schornagel QC, Thijs-Visser MF, van Alphen RJ, Struik LEM, Zuetenhorst HJM, Mathijssen RHJ, Koolen SLW. Therapeutic Drug Monitoring of Endoxifen for Tamoxifen Precision Dosing: Feasible in Patients with Hormone-Sensitive Breast Cancer. Clin Pharmacokinet. 2022 Apr;61(4):527-537. doi: 10.1007/s40262-021-01077-z. Epub 2021 Nov 17. PMID 34786650
- [Background] Sanchez-Spitman A, Dezentje V, Swen J, Moes DJAR, Bohringer S, Batman E, van Druten E, Smorenburg C, van Bochove A, Zeillemaker A, Jongen L, Los M, Neven P, Gelderblom H, Guchelaar HJ. Tamoxifen Pharmacogenetics and Metabolism: Results From the Prospective CYPTAM Study. J Clin Oncol. 2019 Mar 10;37(8):636-646. doi: 10.1200/JCO.18.00307. Epub 2019 Jan 24. PMID 30676859
- [Background] Lu J, Li H, Guo P, Shen R, Luo Y, Ge Q, Shi W, Li Y, Zhu W. The effect of CYP2D6 *10 polymorphism on adjuvant tamoxifen in Asian breast cancer patients: a meta-analysis. Onco Targets Ther. 2017 Nov 13;10:5429-5437. doi: 10.2147/OTT.S149197. eCollection 2017. PMID 29180876